CLINICAL TRIAL: NCT00638833
Title: Pilot Clinical Trial With Memantine for Cognitive Deficits in Patients With Multiple Sclerosis
Brief Title: Memantine Therapy for Multiple Sclerosis
Acronym: Memantine-MS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unexpected side-effects: reversible and mild to moderate neurological impairment
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 11495A
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-06

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Memantine 30 mg/day
  Interventions: Drug: Memantine
- B (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Memantine — Memantine 30 mg/day (20-10-0)
  Other Names: Ebixa
  Arms: A
Drug: Placebo — Placebo pills
  Arms: B

SUMMARY:
To assess the efficacy of Memantine in improving the cognitive impairment in patients with Multiple Sclerosis (MS)

DETAILED DESCRIPTION:
Memantine is an NMDA receptor antagonist that improves cognitive and behavioural deficits in patients with Alzheimer disease, vascular dementia and mixed dementia. This study is focused in proving the efficacy of Memantine in ameliorating one of the most frequent symptoms of patients with MS which is attention and memory deficits. Memantine is a safe drug in patients with MS and it has been administered to MS patients with pendular nystagmus (Starck et al J Neurol 1997). The study will have the power to detect differences in such clinical question by studying 60 MS patients with cognitive impairment (n=60)) with a crossover design. Indeed, we plan to use a new and powerful surrogate marker such as attention evoked potentials developed in our center. Finally, because there are evidences that Memantine might improve MS outcome by closing the Brain-Blood barrier (which is the best therapeutic target in this disease) (Paul et al J Pharmacol Exp Ther 2002), an exploratory study of its efficacy in preventing new MRI lesions might also be included in the design.

Aims: To assess the efficacy of Memantine in improving the cognitive impairment in patients with Multiple Sclerosis (MS) Primary end-point: to assess the efficacy of Memantine in improving memory deficit in MS patients using the SRT scale

Secondary end-points:

1. To assess the efficacy of Memantine in improving the performance in the individual neuropsychological tests for attention (PASAT3, SDMT, Stroop), executive (Raven, MATTIS) and memory (10/36, SRT), in the neuropsychological global scale BRB-N Z (Sepulcre et al, submitted) in quality of life (SF36), disability (EDSS, MSFC, MSSS) and fatigue (Krupp).
2. to assess the effect of Memantine in attention evoked potentials (EP)
3. to assess the effect of Memantine in clinical course (new relapses, relapse rate, patients free of relapses), disability (EDSS, MSFC, MSSS) and MRI parameters (active lesions: new T2 lesions, change in T2 lesion load, new gadolinium enhancing lesions and global and regional atrophy) in the response to Memantine. MRI study is optional.
4. to identify the predictors of good or bad response to Memantine therapy by using EP as surrogate markers.

Design: double blind, randomize and crossover clinical trial with Memantine compared with placebo in MS patients. Because Memantine have a hal-life of 2 to 4 days period, at the end of the 6 month, patients we will stay 3 weeks without any therapy (placebo or Memantine) in order to washout Memantine in the therapeutic group

ELIGIBILITY:
Inclusion Criteria:

* Patients with MS (McDonald 2002), both sex, age between 18 to 60 years old, all MS subtypes (RR, SP, PP, PR), stable.
* Patients with severe cognitive impairment defined as performing 1.5 SD below control group (matched by age and education) in 2 o more subtests based in our previous study (Sepulcre 2006):

Exclusion Criteria:

* Psychiatric diseases (Cummings) depression (Hamilton >8), drug or alcohol abuse, benzodiazepine therapy or other medical diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-09; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
to assess the efficacy of Memantine in improving memory deficit in MS patients using the SRT scale | 6 months

SECONDARY OUTCOMES:
1. tests for attention (PASAT3, SDMT, Stroop), executive (Raven, MATTIS) and memory (10/36, SRT), quality of life (SF36), and fatigue (Krupp). 2. attention evoked potentials 3. clinical course, disability (EDSS, MSFC, MSSS). | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Villoslada, MD, Principal Investigator — University of Navarra
Locations (1):
- Clinica Universitaria de Navarra, Pamplona, Navarre, Spain

REFERENCES:
- [Background] Sepulcre J, Vanotti S, Hernandez R, Sandoval G, Caceres F, Garcea O, Villoslada P. Cognitive impairment in patients with multiple sclerosis using the Brief Repeatable Battery-Neuropsychology test. Mult Scler. 2006 Apr;12(2):187-95. doi: 10.1191/1352458506ms1258oa. PMID 16629422
- [Derived] Villoslada P, Arrondo G, Sepulcre J, Alegre M, Artieda J. Memantine induces reversible neurologic impairment in patients with MS. Neurology. 2009 May 12;72(19):1630-3. doi: 10.1212/01.wnl.0000342388.73185.80. Epub 2008 Dec 17. PMID 19092106
- See also: web page of the medical center of the University of Navarra — http://www.cun.es